CLINICAL TRIAL: NCT07228780
Title: Impact of Resistance Training With and Without Venous Occlusion on Strength and Function Post Hand Burn
Brief Title: Impact of Resistance Training With and Without Venous Occlusion on Strength and Function Post (Hand Burn)
Acronym: hand burn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Gamal Fouad Eltelemy, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006079
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Hand Burn
Keywords: hand burn-hand grip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (aspirin Group) (Experimental): Resistance exercises with venous occlusion This group will include 17 patients with hand burn who will receive treatment for burn which included: positioning, range of motion, stretch, joint mobilization and strength exercise for hand grip with blood flow restriction3 days per week for 4 weeks
  Interventions: Other: resistance exercise with venous occlusion
- control (Experimental): This group will include 17 patients with hand burn who will receive treatment for burn which included: positioning, range of motion, stretch, joint mobilization and strength exercise for hand grip with blood flow restriction3 days per week for 4 weeks
  Interventions: Other: traditional resistance exercises

INTERVENTIONS:
Other: resistance exercise with venous occlusion — patients with hand burn who will receive conventional treatment for burn which included: positioning, range of motion, stretch, joint mobilization and strength exercise for hand grip for 3 days per week for 4 weeks
  Arms: study group (aspirin Group)
Other: traditional resistance exercises — This group will include 17 patients with hand burn who will receive conventional treatment for burn which included: positioning, range of motion, stretch, joint mobilization and strength exercise for hand grip for 3 days per week for 4 weeks
  Arms: control

SUMMARY:
It will be hypothesized that There is There is no difference between resistance training with and without venous occlusion on hand strength and function post hand burn.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the difference between resistance training with and without venous occlusion on hand strength and function post hand burn.

This study will be designed to evaluate the difference between resistance training with and without venous occlusion on hand strength and function post hand burn.

ELIGIBILITY:
Inclusion Criteria:

* Patients of all age groups and both sexes having less than sixty percent TBSA thermal burns and involves the hand.

  * Patients with second-degree (superficial or deep) burn on the hand.
  * Patients with third-degree burns
  * Patients with complete wound healing
  * Patients without any defects at tendons
  * Patients without burning at cubital fossa (cuff placement)
  * participants were required to have a resting (systolic and diastolic) blood pressure of <140/90 mmHg and a resting heart rate of <90 bpm
  * A decreased grip strength.
  * Patients without cognitive impairments and actively cooperating with treatment and measurements

Exclusion Criteria:

* Any patient who has previous injury or congenital deformity of the hand with restricted hand function.
* Resting systolic BP (BP) <140 mmHg and/or diastolic BP< 90 mmHg
* Self-reported cardiovascular, metabolic, or pulmonary conditions or signs and symptoms suggestive of these diseases
* Associated injuries affecting participation in exercise training, including fracture, amputation, acquired brain injury or peripheral neural injury or any pre-existing medical condition which may affect exercise participation.
* patients that had fourth degree burns
* patients that had first degree burns
* Patients with burn at cubital fossa (cuff placement)
* Patients without complete wound healing
* patient who is taking medications that affect hemodynamic responses
* Patients with severe hand burns leading to muscle and tendon damage, or those who have undergone finger amputation surgery
* Patients who were not compliant for following up for at least once a month following discharge from hospital.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
hand grip strength | twice first before beginning treatment from day 1 of treatment second after complete treatment after 1 month Assessment will be for 1 minute For assessment hand grip strength
  Hand grip will be assessed by digital Hand Dynamometer

SECONDARY OUTCOMES:
upper limb function | twice first pre treatment at 1 day for almost 5 minutes to assess all functions of upper limb function second after complete treatment after 1 month to assess upper limb function after treatment for 5 minutes
  Function of hand will be assessed by quick disabilities of arm, shoulder and hand questionnaire which asks patient about symptoms as well as ability to perform certain activities This scale which which assess upper limb function and high score means high disability and bad results and low score means low disability and good results

IPD SHARING:
Plan to Share IPD: No
it is considered privacy of patients and privacy of my research

REFERENCES:
- [Result] Araujo, B. F., do Nascimento, C. M., Busarello, F. O., Moreira, N. B., Baroni, M. P., de Carvalho, A. R., & Bertolini, G. R. F. (2012). Assessment of handgrip strength after neural mobilization. Revista Brasileira de Medicina do Esporte, 18(4), 242-245.
- [Result] Ahmed, A. M., Hassan, Y. S., Azer, S. Z., & Abd EL-All, H. A. E. R. (2019). Effect of range of motion exercise program on improving upper-arm region joints function for burned patients. Assiut Scientific Nursing Journal, 7(19), 61-69.
- [Result] Watzinger N, Hecker A, Petschnig D, Tran J, Glantschnig C, Moshammer M, Pignet AL, Ellersdorfer AM, Kamolz LP. Long-Term Functional Outcomes after Hand Burns: A Monocentric Controlled Cohort Study. J Clin Med. 2024 Jun 15;13(12):3509. doi: 10.3390/jcm13123509. PMID 38930038
- [Result] Watson R, Sullivan B, Stone A, Jacobs C, Malone T, Heebner N, Noehren B. Blood Flow Restriction Therapy: An Evidence-Based Approach to Postoperative Rehabilitation. JBJS Rev. 2022 Oct 3;10(10). doi: 10.2106/JBJS.RVW.22.00062. eCollection 2022 Oct 1. PMID 36191086
- [Result] Tehreem, Z., Kazmi, Y., Khalid, M. U., Mansha, H., Hassan, M., & Majeed, R. (2022). Comparison of soft tissue mobilization versus static stretching in post-burn contractures at elbow and wrist, A pilot study. Journal of University Medical & Dental College, 13(3), 408-411.
- [Result] Serghiou M, Cowan A, Whitehead C. Rehabilitation after a burn injury. Clin Plast Surg. 2009 Oct;36(4):675-86. doi: 10.1016/j.cps.2009.05.008. PMID 19793561
- [Result] Schoenfeld BJ. The mechanisms of muscle hypertrophy and their application to resistance training. J Strength Cond Res. 2010 Oct;24(10):2857-72. doi: 10.1519/JSC.0b013e3181e840f3. PMID 20847704
- [Result] Salwa, F., KHATTAB, A. S., MOHAMMED, M. M., & NASER, M. A. (2020). Validity and reliability of the Arabic version of the quick-dash questionnaire for upper extremity disorders. The Medical Journal of Cairo University, 88(December), 2037-2043
- [Result] Reina-Ruiz AJ, Martinez-Cal J, Molina-Torres G, Romero-Galisteo RP, Galan-Mercant A, Carrasco-Vega E, Gonzalez-Sanchez M. Effectiveness of Blood Flow Restriction on Functionality, Quality of Life and Pain in Patients with Neuromusculoskeletal Pathologies: A Systematic Review. Int J Environ Res Public Health. 2023 Jan 12;20(2):1401. doi: 10.3390/ijerph20021401. PMID 36674158
- [Result] Prolonge, R. (2022). Hand and Wrist Mobilizations. In: Mesplié, G. (eds) Hand and Wrist Therapy. Springer, Cham. https://doi.org/10.1007/978-3-030-94942-6_5
- [Result] Procter F. Rehabilitation of the burn patient. Indian J Plast Surg. 2010 Sep;43(Suppl):S101-13. doi: 10.4103/0970-0358.70730. PMID 21321643
- [Result] Perera, A. D., Perera, C., & Karunanayake, A. L. (2017). Effectiveness of early stretching exercises for range of motion in the shoulder joint and quality of functional recovery in patients with burns-a randomized control trial.
- [Result] Mohammadabadi, H. D., Azizi, S., Dadarkhah, A., & Soltani, Z. R. (2018). Evaluation of effectiveness of the wrist mobilization compared with local corticosteroid injection in treatment of moderate carpal tunnel syndrome. Annals of Military and Health Sciences Research, 16(2), e83335.
- [Result] Machek, S. B., Harris, D. R., Heileson, J. L., Wilburn, D. T., Forsse, J. S., & Willoughby, D. S. (2023). Impacts of varying blood flow restriction cuff size and material on arterial, venous and calf muscle pump-mediated blood flow. Oxygen, 3(2), 190-202
- [Result] Kara S, Seyhan N, Oksuz S. Effectiveness of early rehabilitation in hand burns. Ulus Travma Acil Cerrahi Derg. 2023 Jun;29(6):691-697. doi: 10.14744/tjtes.2023.22780. PMID 37278077
- [Result] Joseph, S. (2022). The effective management and outcome of hand burns. *Journal of Clinical Research and Reports, 10*(1). https://doi.org/10.31579/2690-1919/213
- [Result] Hornikel B, Saffold KS, Esco MR, Mota JA, Fedewa MV, Wind SA, Adams TL, Winchester LJ. Acute Responses to High-Intensity Back Squats with Bilateral Blood Flow Restriction. Int J Environ Res Public Health. 2023 Feb 17;20(4):3555. doi: 10.3390/ijerph20043555. PMID 36834246
- [Result] Heiser R, O'Brien VH, Schwartz DA. The use of joint mobilization to improve clinical outcomes in hand therapy: a systematic review of the literature. J Hand Ther. 2013 Oct-Dec;26(4):297-311; quiz 311. doi: 10.1016/j.jht.2013.07.004. Epub 2013 Sep 14. PMID 24044954
- [Result] Gün, N., Kavlak, B., Sarı, Z., & Yurdalan, S. U. (2023). The effect of neural mobilization on muscle strength, reaction time, and pain threshold. *Turkish Journal of Science and Health, 4*(2), 155-162. https://doi.org/10.51972/tfsd.1233200
- [Result] Gittings P, Salet M, Burrows S, Ruettermann M, Wood FM, Edgar D. Grip and Muscle Strength Dynamometry Are Reliable and Valid in Patients With Unhealed Minor Burn Wounds. J Burn Care Res. 2016 Nov/Dec;37(6):388-396. doi: 10.1097/BCR.0000000000000414. PMID 27606549
- [Result] Franz A, Ji S, Froschen FS, Kerstin M, Wahl P, Behringer M. Effects of low-load blood flow restriction on the venous system in comparison to traditional low-load and high-load exercises. Front Physiol. 2023 Dec 15;14:1285462. doi: 10.3389/fphys.2023.1285462. eCollection 2023. PMID 38162828
- [Result] Franz A, Ji S, Bittersohl B, Zilkens C, Behringer M. Impact of a Six-Week Prehabilitation With Blood-Flow Restriction Training on Pre- and Postoperative Skeletal Muscle Mass and Strength in Patients Receiving Primary Total Knee Arthroplasty. Front Physiol. 2022 Jun 14;13:881484. doi: 10.3389/fphys.2022.881484. eCollection 2022. PMID 35774280
- [Result] 15. Filippou, S., Iakovidis, P., Lytras, D., Kasimis, K., Solomonidou, F., & Kopsidas, C. (2023). Hemodynamic Responses to a Handgrip Exercise Session, with and without Blood Flow Restriction, in Healthy Volunteers. Physiologia, 3(2), 259-271.
- [Result] Fernandes DZ, Weber VMR, da Silva MPA, de Lima Stavinski NG, de Oliveira LEC, Casoto Tracz EH, Ferreira SA, da Silva DF, Queiroga MR. EFFECTS OF BLOOD FLOW RESTRICTION TRAINING ON HANDGRIP STRENGTH AND MUSCULAR VOLUME OF YOUNG WOMEN. Int J Sports Phys Ther. 2020 Dec;15(6):901-909. doi: 10.26603/ijspt20200901. PMID 33344006
- [Result] Edger-Lacoursiere Z, Deziel E, Nedelec B. Rehabilitation interventions after hand burn injury in adults: A systematic review. Burns. 2023 May;49(3):516-553. doi: 10.1016/j.burns.2022.05.005. Epub 2022 May 14. PMID 35662480
- [Result] Credeur DP, Hollis BC, Welsch MA. Effects of handgrip training with venous restriction on brachial artery vasodilation. Med Sci Sports Exerc. 2010 Jul;42(7):1296-302. doi: 10.1249/MSS.0b013e3181ca7b06. PMID 20019641
- [Result] 10. Costa, C. R. M., Dos-Santos, R. C., Paula, W. V., Ribeiro, W. M. V., & Silveira, A. L. B. (2017). Acute static muscle stretching improves manual dexterity in young men. *MedicalExpress (São Paulo, online), 4*(3), M170306. https://doi.org/10.5935/MedicalExpress.2017.03.06
- [Result] 8. Cerqueira, M. S., Pereira, R., Mesquita, G. N. D., Rocha, T., & Moura Filho, A. G. D. (2019). Rate of force development to evaluate the neuromuscular fatigue and recovery after an intermittent isometric handgrip task with different blood flow restriction conditions. Motriz: Revista de Educação Física, 25(1), e1019123.
- [Result] Bryant J, Cooper DJ, Peters DM, Cook MD. The Effects of Static Stretching Intensity on Range of Motion and Strength: A Systematic Review. J Funct Morphol Kinesiol. 2023 Mar 24;8(2):37. doi: 10.3390/jfmk8020037. PMID 37092369
- [Result] Bond CW, Hackney KJ, Brown SL, Noonan BC. Blood Flow Restriction Resistance Exercise as a Rehabilitation Modality Following Orthopaedic Surgery: A Review of Venous Thromboembolism Risk. J Orthop Sports Phys Ther. 2019 Jan;49(1):17-27. doi: 10.2519/jospt.2019.8375. Epub 2018 Sep 12. PMID 30208794
- [Result] Davies TW, Kelly E, van Gassel RJJ, van de Poll MCG, Gunst J, Casaer MP, Christopher KB, Preiser JC, Hill A, Gundogan K, Reintam-Blaser A, Rousseau AF, Hodgson C, Needham DM, Schaller SJ, McClelland T, Pilkington JJ, Sevin CM, Wischmeyer PE, Lee ZY, Govil D, Chapple L, Denehy L, Montejo-Gonzalez JC, Taylor B, Bear DE, Pearse RM, McNelly A, Prowle J, Puthucheary ZA. A systematic review and meta-analysis of the clinimetric properties of the core outcome measurement instruments for clinical effectiveness trials of nutritional and metabolic interventions in critical illness (CONCISE). Crit Care. 2023 Nov 20;27(1):450. doi: 10.1186/s13054-023-04729-7. PMID 37986015
- [Result] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Result] Araujo CG, Duarte CV, Goncalves Fde A, Medeiros HB, Lemos FA, Gouvea AL. Hemodynamic responses to an isometric handgrip training protocol. Arq Bras Cardiol. 2011 Nov;97(5):413-9. doi: 10.1590/s0066-782x2011005000102. Epub 2011 Oct 21. English, Portuguese. PMID 22011802